CLINICAL TRIAL: NCT06272084
Title: Analysis of TPE Treatments With multiFiltratePRO
Acronym: TPEopt
Status: Recruiting | Type: Observational
Sponsor: Fresenius Medical Care Deutschland GmbH (Industry)
Collaborators: X-act Cologne Clinical Research GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: CRRT-TPE-01-DE
Record Dates: First submitted 2024-02-05; First posted 2024-02-22 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Autoimmune Diseases
Keywords: Therapeutical Plasma Exchange; ASFA Guideline
MeSH Terms: conditions — Autoimmune Diseases | interventions — Plasma Exchange

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- TPE Treatments: Patients with indication for TPE treatment according to American Society for Apheresis (ASFA) guideline
  Interventions: Device: Therapeutic Plasma Exchange (TPE) option of multiFiltratePRO

INTERVENTIONS:
Device: Therapeutic Plasma Exchange (TPE) option of multiFiltratePRO — Retrospective Data Analysis of TPE treatments with multiFiltratePRO

SUMMARY:
Analysis of therapeutic plasma exchange (TPE) treatments to assess the performance of the TPE mode of multiFiltratePRO based on the successful exchange of plasma from whole blood. The multiFiltratePRO is a device for extracorporeal blood purification treatments.

DETAILED DESCRIPTION:
The study is a retrospective, open, non-comparative, multi-centric PMCF study. The investigational device has CE approval. The investigation involves the retrospective collection of treatment data for the TPE treatment mode from the medical records. No further control treatments will be investigated in this one-arm design. The design is considered to be appropriate to reflect daily clinical practice and to contribute to empirical evidence of performance of the TPE mode of the multiFiltratePRO system.

The site will document the treatment data of patients with an indication for the TPE treatment who had been treated with the investigational devices under the TPE treatment mode between 2019 and October 2023 in chronological order.

ELIGIBILITY:
Inclusion Criteria:

* Body weight ≥40kg irrespective of the age
* Patients with indication for TPE treatment according to ASFA guideline
* Patients have been treated with TPE between January 2019 and October 2023
* Availability of at least 50% of the parameters to be documented for the patient

Exclusion Criteria:

* Participation in an interventional clinical study during the retrospectively collected TPE treatment data
* Previous documentation within this study
* Simultaneous use of another filter for additional therapy form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with indication for TPE treatment according to ASFA (American Society for Apheresis) guideline treated with TPE between January 2019 and October 2023.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-05-22 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Total amount of exchange plasma (prescribed vs achieved exchange volume) | through study completion, an average of 1 year
  Statistical analysis is performed on retrospective data (Treatments between 2019 and October 2023). Primary goal of the study is to prove that the prescribed therapeutic plasma exchange rate during treatment was achieved in > 70% of treatments and therefore was in alignment with current guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Büttner, Dr. med., Principal Investigator — Klinikum Aschaffenburg-Alzenau
Locations (3):
- Germany (3):
  - Klinikum Aschaffenburg-Alzenau, Aschaffenburg, Bavaria
  - Universitätsklinikum Würzburg, Würzburg, Bavaria
  - Charité-Universitätsmedizin Berlin, Berlin, State of Berlin

IPD SHARING:
Plan to Share IPD: No